CLINICAL TRIAL: NCT03081832
Title: Long Term Evaluation of Infants Aged From 3 to 4 Years Old Included in the Ancient Study (Repeated Administrations of Oxytocin in Infants With Prader Willi Syndrome Aged From 0 to 6 Months) and Comparison With Not Treated and Age-matched Prader Willi Syndrome Infants (OT2SUITE)
Brief Title: Follow-up of Prader Willi Syndrome Infants Treated by Oxytocin and Comparison With Not-treated Infants.
Acronym: OT2SUITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/16/8407; 2016-A01348-43 (Other: ID-RCB)
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi; Oxytocin; Communication skills; Oral skills; Brain activity; Hormonal disease
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Groups of children with Prader Willi Syndrome treated by oxytocin for 7 days during their first 6 months of life.
  Interventions: Drug: Oxytocin
- Control (Experimental): Groups of children with Prader Willi Syndrome not treated by oxytocin for 7 days during their first 6 months of life.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Oxytocin — Infant included in the ancient study (repeated administrations of oxytocin in infants with Prader Willi Syndrome aged from 0 to 6 months)
  Arms: Oxytocin
Other: Control — Not treated.
  Arms: Control

SUMMARY:
The objective of this study is to collect data on tolerance and effects of early treatment with oxytocin in children with Prader Willi Syndrome aged from 3 to 4 years and to compare these infants with not treated age-matched infants with Prader Willi Syndrome.

DETAILED DESCRIPTION:
In accordance with recommendations of regulatory authorities, we want to collect long term data of patients treated with oxytocin before the age of 6 months. Moreover clinical observations of these infants support long term effects on communication skills, global development and behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Infants with Prader Willi Syndrome (genetic diagnosis confirmed)
* For treated group : infant included in the ancient study
* For not treated group: infant never treated with oxytocin

Exclusion Criteria:

* Subject involved in another search including an exclusion period still in progress at the time of inclusion.
* Impossibility to give parents or legal guardian informed information
* No coverage by a Social Security scheme
* Refusal of parents or legal representative to sign consent.

If a patient has a contraindication to Magnetic resonance imaging, it may be included in the study but Magnetic resonance imaging will not be performed.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of communication skills. | Day 1
  Assessed by Vineland-II scale.

SECONDARY OUTCOMES:
Evaluation of adaptative behavior composite and 3 domains : "Daily living skills", "Socialization", "Motor skills". | Day 1
  Assessed by Vineland-II scale.
Evaluation of behavioral troubles. | Day 1
  Assessed by Child Behaviour Check List questionnaire.
Evaluation of global development. | Day 2 and 3
  Assessed by Bayley Scales of Infant and Toddler Development.
Evaluation of orality and eating behaviour. | Day 2
  Assessed by:
  * A questionnaire on eating behavior.
  * An oral evaluation, which combines a clinical examination carried out by the reference center physician, and the assessment of eating behavior during the meal.
  * The fluoroscopy of swallowing.
Evaluation of brain activity. | Day 3
  Assessed by a morphological Magnetic resonance imaging, a resting functional Magnetic resonance imaging.
Evaluation of plasma levels of ghrelin and other peptides involved in feeding behaviour or energy metabolism. | Day 1
  Circulating levels of acylated and non-acylated ghrelin and some peptides and neuropeptides involved in appetite regulation (leptin, cortisol, insulin, Glucagon like peptide-1, pancreatic polypeptide, orexin A, alpha-melanocyte stimulating hormone...).

CONTACTS AND LOCATIONS:
Overall Officials: Maïthé Tauber, Pr, Principal Investigator — Centre de référence du syndrome de Prader-Willi- CHU Toulouse
Locations (1):
- Centre de référence du syndrome de Prader-Willi Hôpital des Enfants, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amico JA, Vollmer RR, Cai HM, Miedlar JA, Rinaman L. Enhanced initial and sustained intake of sucrose solution in mice with an oxytocin gene deletion. Am J Physiol Regul Integr Comp Physiol. 2005 Dec;289(6):R1798-806. doi: 10.1152/ajpregu.00558.2005. Epub 2005 Sep 8. PMID 16150836
- [Background] Arletti R, Benelli A, Bertolini A. Oxytocin inhibits food and fluid intake in rats. Physiol Behav. 1990 Dec;48(6):825-30. doi: 10.1016/0031-9384(90)90234-u. PMID 2087513
- [Background] Billings LB, Spero JA, Vollmer RR, Amico JA. Oxytocin null mice ingest enhanced amounts of sweet solutions during light and dark cycles and during repeated shaker stress. Behav Brain Res. 2006 Jul 15;171(1):134-41. doi: 10.1016/j.bbr.2006.03.028. Epub 2006 May 4. PMID 16677726
- [Background] Bittel DC, Kibiryeva N, Sell SM, Strong TV, Butler MG. Whole genome microarray analysis of gene expression in Prader-Willi syndrome. Am J Med Genet A. 2007 Mar 1;143A(5):430-42. doi: 10.1002/ajmg.a.31606. PMID 17236194
- [Background] Dykens EM, Lee E, Roof E. Prader-Willi syndrome and autism spectrum disorders: an evolving story. J Neurodev Disord. 2011 Sep;3(3):225-37. doi: 10.1007/s11689-011-9092-5. Epub 2011 Aug 20. PMID 21858456
- [Background] Dykens EM, Maxwell MA, Pantino E, Kossler R, Roof E. Assessment of hyperphagia in Prader-Willi syndrome. Obesity (Silver Spring). 2007 Jul;15(7):1816-26. doi: 10.1038/oby.2007.216. PMID 17636101
- [Background] Dykens EM, Roof E, Hunt-Hawkins H. Cognitive and adaptive advantages of growth hormone treatment in children with Prader-Willi syndrome. J Child Psychol Psychiatry. 2017 Jan;58(1):64-74. doi: 10.1111/jcpp.12601. Epub 2016 Aug 2. PMID 27481444
- [Background] Goldstone AP, Holland AJ, Butler JV, Whittington JE. Appetite hormones and the transition to hyperphagia in children with Prader-Willi syndrome. Int J Obes (Lond). 2012 Dec;36(12):1564-70. doi: 10.1038/ijo.2011.274. Epub 2012 Jan 24. PMID 22270375
- [Background] Guastella AJ, Einfeld SL, Gray KM, Rinehart NJ, Tonge BJ, Lambert TJ, Hickie IB. Intranasal oxytocin improves emotion recognition for youth with autism spectrum disorders. Biol Psychiatry. 2010 Apr 1;67(7):692-4. doi: 10.1016/j.biopsych.2009.09.020. Epub 2009 Nov 7. PMID 19897177
- [Background] Hall SS, Lightbody AA, McCarthy BE, Parker KJ, Reiss AL. Effects of intranasal oxytocin on social anxiety in males with fragile X syndrome. Psychoneuroendocrinology. 2012 Apr;37(4):509-18. doi: 10.1016/j.psyneuen.2011.07.020. Epub 2011 Aug 20. PMID 21862226
- [Background] Kosfeld M, Heinrichs M, Zak PJ, Fischbacher U, Fehr E. Oxytocin increases trust in humans. Nature. 2005 Jun 2;435(7042):673-6. doi: 10.1038/nature03701. PMID 15931222
- [Background] Lischke A, Gamer M, Berger C, Grossmann A, Hauenstein K, Heinrichs M, Herpertz SC, Domes G. Oxytocin increases amygdala reactivity to threatening scenes in females. Psychoneuroendocrinology. 2012 Sep;37(9):1431-8. doi: 10.1016/j.psyneuen.2012.01.011. Epub 2012 Feb 23. PMID 22365820
- [Background] McDonald NA, Kuzmiski JB, Naderi N, Schwab Y, Pittman QJ. Endogenous modulators of synaptic transmission: cannabinoid regulation in the supraoptic nucleus. Prog Brain Res. 2008;170:129-36. doi: 10.1016/S0079-6123(08)00412-3. PMID 18655878
- [Background] Meziane H, Schaller F, Bauer S, Villard C, Matarazzo V, Riet F, Guillon G, Lafitte D, Desarmenien MG, Tauber M, Muscatelli F. An Early Postnatal Oxytocin Treatment Prevents Social and Learning Deficits in Adult Mice Deficient for Magel2, a Gene Involved in Prader-Willi Syndrome and Autism. Biol Psychiatry. 2015 Jul 15;78(2):85-94. doi: 10.1016/j.biopsych.2014.11.010. Epub 2014 Nov 20. PMID 25599930
- [Background] Miller JL, Lynn CH, Driscoll DC, Goldstone AP, Gold JA, Kimonis V, Dykens E, Butler MG, Shuster JJ, Driscoll DJ. Nutritional phases in Prader-Willi syndrome. Am J Med Genet A. 2011 May;155A(5):1040-9. doi: 10.1002/ajmg.a.33951. Epub 2011 Apr 4. PMID 21465655
- [Background] Salles J, Strelnikov K, Carine M, Denise T, Laurier V, Molinas C, Tauber M, Barone P. Deficits in voice and multisensory processing in patients with Prader-Willi syndrome. Neuropsychologia. 2016 May;85:137-47. doi: 10.1016/j.neuropsychologia.2016.03.015. Epub 2016 Mar 16. PMID 26994593
- [Background] Schaller F, Watrin F, Sturny R, Massacrier A, Szepetowski P, Muscatelli F. A single postnatal injection of oxytocin rescues the lethal feeding behaviour in mouse newborns deficient for the imprinted Magel2 gene. Hum Mol Genet. 2010 Dec 15;19(24):4895-905. doi: 10.1093/hmg/ddq424. Epub 2010 Sep 28. PMID 20876615
- [Background] Skokauskas N, Sweeny E, Meehan J, Gallagher L. Mental health problems in children with prader-willi syndrome. J Can Acad Child Adolesc Psychiatry. 2012 Aug;21(3):194-203. PMID 22876265
- [Background] Swaab DF, Purba JS, Hofman MA. Alterations in the hypothalamic paraventricular nucleus and its oxytocin neurons (putative satiety cells) in Prader-Willi syndrome: a study of five cases. J Clin Endocrinol Metab. 1995 Feb;80(2):573-9. doi: 10.1210/jcem.80.2.7852523.
- [Background] van Lieshout CF, de Meyer RE, Curfs LM, Koot HM, Fryns JP. Problem behaviors and personality of children and adolescents with Prader-Willi syndrome. J Pediatr Psychol. 1998 Apr;23(2):111-20. doi: 10.1093/jpepsy/23.2.111. PMID 9585637
- [Derived] Valette M, Diene G, Glattard M, Cortadellas J, Molinas C, Faye S, Benvegnu G, Boulanouar K, Payoux P, Salles JP, Arnaud C, Cabal S, Tauber M. Early oxytocin treatment in infants with Prader-Willi syndrome is safe and is associated with better endocrine, metabolic and behavioral outcomes. Orphanet J Rare Dis. 2025 Mar 1;20(1):96. doi: 10.1186/s13023-025-03560-3. PMID 40025514